CLINICAL TRIAL: NCT03851627
Title: 52 Week RCT to Investigate the Effect of Testosterone Undecanoate vs Placebo on Intrahepatic Fat Content in Obese/Overweight Men With T2DM/Prediabetes and Hypogonadism and Subsequent 108 Week Open Label Phase to Investigate Effects on Cardiometabolic Parameters
Brief Title: Effects of Testosterone Undecanoate vs Placebo on Intrahepatic Fat Content in Overweight/Obese Men With T2DM or Prediabetes and Hypogonadism
Acronym: Test2Func
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandra Kautzky-Willer (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Alexandra Kautzky-Willer, Head of Department of Endocrinology, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: T2F12017; 2017-001611-37 (EudraCT Number)
Record Dates: First submitted 2019-01-14; First posted 2019-02-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fatty Liver; Overweight/Obesity; Prediabetes/Type2 Diabetes Mellitus; Hypogonadism, Male
MeSH Terms: conditions — Fatty Liver; Overweight; Obesity; Prediabetic State; Eunuchism | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone undecanoate (Active Comparator): intramuscular Testosterone undecanoate 1000mg/4ml
  Interventions: Drug: Testosterone Undecanoate
- Testosterone like Placebo (Placebo Comparator): intramuscular Testosterone undecanoate like Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Undecanoate — 1000mg/4ml i.m. initial, after 6 weeks, every 10 weeks thereafter
  Other Names: Nebido
  Arms: Testosterone undecanoate
Drug: Placebo — Placebo Arm
  Other Names: oily solution, Nebido like Placebo
  Arms: Testosterone like Placebo

SUMMARY:
The epidemics of obesity, MeTSy, T2DM and CVD are increasing worldwide. Non-alcoholic fatty liver disease (NAFLD) is becoming recognized as a condition possibly involved in the pathogenesis of these diseases. The prevailing hypothesis for NAFLD pathogenesis is the 'two-hit' model, with insulin resistance and hyperinsulinemia playing essential roles, which have a plethora of effects on hepatic lipid metabolism and can lead to accumulation of triglycerides in hepatocytes. Accepted treatment for NAFLD is lifestyle modifications. Sex hormones might be relevant in T2DM development and treatment. Low testosterone (T) has deteriorating effects on glucose levels, and aggravates in obesity as aromatization of T is enhanced. T deficiency is related to increases of visceral fat accumulation and associated with development of NAFLD. T replacement might be a successful way in hypogonadism to treat obesity and counteract progression of MEtSy,T2DM or CVD driven by visceral fat accumulation or NAFLD.

Primary Objective To investigate the effects on hepatic lipid content reduction of a therapy with Testosterone undecanoate 1000mg compared to placebo given for 52 weeks in patients with type 2 diabetes mellitus and hypogonadism.

DETAILED DESCRIPTION:
Background The epidemics of obesity, metabolic syndrome, type 2 diabetes, and atherosclerosis are increasing worldwide. Non-alcoholic fatty liver disease (NAFLD), for a long time unnoted in the metabolic field, is becoming recognized as a condition possibly involved in the pathogenesis of these diseases. Support for this hypothesis emerges from studies revealing that NAFLD precedes the manifestation of the metabolic derangements. NAFLD includes the whole spectrum from non-evolutive simple steatosis to progressive non-alcoholic steatohepatitis (NASH) with/without cirrhosis and hepatocellular carcinoma in individuals without relevant alcohol consumption. NAFLD is a relevant issue in public health owing to its' epidemiologic burden. It represents the most common chronic liver disease in the general population and is expected to increase in the future as a result of an ageing population, the improving control of other major causes of chronic liver disease and the epidemics of obesity and diabetes. The prevalence of NAFLD varies according to age, gender and ethnicity. In the general population, the prevalence of NAFLD is about 25% and the incidence is of two new cases/100 people/year. 2-3% of individuals in the general population will suffer from NASH. Furthermore, up to 15-20% of patients with NASH may develop cirrhosis and 30-40%of these patients who develop cirrhosis may suffer from liver-related mortality. NAFLD is tightly associated with the metabolic syndrome. The metabolic syndrome is a condition characterized by a cluster of alterations including glucose intolerance/ insulin resistance, abdominal obesity, atherogenic dyslipidemia (low concentrations of high density lipoprotein- cholesterol and high concentrations of triglycerides), elevated blood pressure, a proinflammatory and a prothrombotic state. It increases morbidity and mortality, especially due to cardiovascular disease. The prevailing hypothesis for NAFLD pathogenesis is the 'two-hit' model, with insulin resistance and hyperinsulinemia playing essential roles. Insulin resistance and hyperinsulinemia have a plethora of effects on hepatic lipid metabolism and can lead to accumulation of excess triglycerides in hepatocytes. The progression to NASH entails a 'second hit', which is believed to be due to oxidative stress, upregulation of inflammatory mediators, and dysregulated apoptosis, resulting in inflammation (producing NASH) and fibrosis. Currently, the only accepted treatment for NAFLD regardless of stage is lifestyle modifications. These include weight loss by a combination of decreased caloric intake and increased physical activity.

Study rationale Many patients worldwide are suffering from type 2 diabetes with steeply rising numbers predicted for the next decades. Although much progress can be seen in the field of diabetic research and new treatment modalities, new approaches have to be found to cure the disease and underlying risk factors. As men and women show sex specific differences especially in risk factors of T2DM, a sex- and gender-sensitive approach might be considered. Sex hormones might play an important role in the development and possibly the treatment of T2DM. In women higher but in men lower than normal testosterone concentrations predispose for a higher diabetes risk making evident that sex hormones and sex hormone equilibrium are relevant in disease progression. Especially in men low testosterone levels have deteriorating effects on glucose levels, which is aggravated in obesity as aromatization of testosterone to estrogen is enhanced. Due to this mechanism changes in energy homeostasis are reported which lead to changes in lipid accumulation, as described for visceral obesity. Testosterone deficiency is related to increases of visceral fat accumulation. Furthermore testosterone deficiency is associated with the development of non alcoholic fatty liver disease (NAFLD), a well known risk factor for progression of metabolic syndrome (MEtSy), T2DM and cardiovascular disease. Thus, testosterone replacement might be a successful way in hypogonadal men to treat obesity and counteract the further progression of MEtSy, T2DM or cardiovascular disease mainly driven by visceral fat accumulation and NAFLD and are able to improve quality of life.

Testosterone and changes in metabolism:

Whether low testosterone levels have direct effects on hyperglycaemia or testosterone deficiency is caused by chronic diseases such as type 2 diabetes is not yet fully understood and needs further clarification.

Studies are showing that the link between hypogonadism and the metabolic syndrome is bidirectional. On the one hand MetSy and obesity are associated with a higher risk of hypogonadism in the future but on the other hand low testosterone levels and SHBG levels are strong predictors for the development of MetSy and T2DM. It is further hypothesized that hypoandrogenism is an early marker for disturbances in glucose metabolism. Many studies proved that low testosterone levels may aggravate hyperglycaemia and also may deteriorate other metabolic parameters such as insulin levels and sensitivity, lipid levels, hepatic, myocardial and visceral fat content or body composition in general. Just recently the ADA recommends to test for testosterone deficiency (morning testosterone levels) in all men with T2DM with symptoms or signs of hypogonadism, which are decreased sexual desire or erectile dysfunction.

Treatment in asymptomatic men is controversial. Supplementation of testosterone in diabetic men with hypogonadism was reported to increase insulin sensitivity and to significantly reduce HbA1c, which was also reported in a long time observational study including men with T2DM with an amelioration of glycemic control as well as other cardiovascular and cardiometabolic parameters. Furthermore, total and LDL cholesterol, as well as lipoprotein a were lowered, and body composition, libido, and sexual function improved, whereas frequencies of adverse events (AEs) or serious AEs between groups were comparable after 6 months of transdermal testosterone application. These results were corroborated by a systematic review including five RCTs with 350 diabetic hypogonadal men showing improvements in fasting glucose, fasting insulin, HbA1c and triglyceride levels. In a recent study depression was found to have confounding effects with alleviated success in reduction in waist circumference, weight, and body mass index as well as improvements in glycaemic control in men with psychiatric disorders. Testosterone is an important regulator of central and peripheral adipose tissue and shows many inhibitory effects such as triglyceride uptake in fat tissue or lipoprotein lipase activity, as well as a higher lipolytic activity triggered by β-adrenergic receptors. An RCT found that in men with hypogonadism subcutaneous fat mass decreases, lean mass and insulin sensitivity increase and the expression of insulin signaling genes is upregulated after testosterone treatment. Furthermore, inflammatory parameters as well as FFA decrease after testosterone treatment. Interestingly in this study a decrease in hepatic lipids in the treatment group was found, which was not significant in a 24 weeks treatment period. However, treatment groups were inhomogenous regarding baseline hepatic lipid content, the lipid content was relatively low for a collective of subjects with T2DM and the treatment period was relatively short. Another recent RCT found significant reductions in HOMA-IR, HbA1c by 0.94 +- 0.88% and an increase in flow-mediated dilatation, which indicates improved endothelial function in a hypogonadal male population with obesity and diabetes.

Testosterone and cardiovascular risk:

The influence of testosterone on cardiovascular risk factors is not well investigated as prospective data are widely missing but evidence shows that testosterone application in men does not increase cardiovascular risk. Furthermore androgen deficiency is associated with a higher risk in cardiovascular mortality. Recent epidemiological data suspect testosterone replacement therapy to increase cardiovascular risk. However, FDA experts find that data is insufficient to make clear suggestions and that there is a need for clinical trials assessing safety of testosterone replacement in people at high risk for cardiovascular risk, like older men, men with T2DM or obesity. After this FDA statement a retrospectively assessed observational study with over 80000 male veterans with documented low total testosterone levels was published reporting a reduction of all cause mortality, myocardial infarction and stroke in men with testosterone replacement therapy. A reduction of MACE was also reported in a further study in male subjects with low testosterone levels substituted to normal levels compared to those with persistent low levels. Men with high testosterone levels had similar MACE risk but a trend for higher stroke risk.

Especially in an obese population with T2DM and hypogonadism the mortality and morbidity caused by coronary artery disease is expected to be high, as CAD is the leading cause of death in subjects with T2DM and often progresses asymptomatic until an infarction or sudden cardiac death occur. Recent conducted MPI (=myocardial perfusion imaging) studies in T2DM patients have shown higher prevalence of abnormal MPI, with more extensive ischemia, compared with subjects without T2DM. The DIAD trial did not show any benefit in prevention of cardiac events comparing MPI screening at regular intervals with a non-screened diabetic population up to nearly 5 years. However, it remains uncertain whether asymptomatic patients with type 2 diabetes benefit from revascularization after the identification of inducible ischemia, as was suggested in a prior retrospective database analysis and a small randomized pilot study. Currently in obese men with hypogonadism and T2DM it is largely unknown whether testosterone replacement has any effects on cardiac perfusion. According to appropriate use criteria (AUC) for the detection a risk assessment of stable ischemic heart disease MPI is a potential diagnostic method to detect CHD at stages of high global coronary artery disease risk [42]. According to NCEP ATP III criteria, the recommended tool of the AUC, the patient collective of TEST2FUNC featuring male subjects with hypogonadism, diabetes mellitus, overweight/obesity, hypertension and dyslipidemia are at high risk for coronary heart disease, as diabetes is seen as a CHD risk equivalent and confers to a high risk of new CHD within 10 years.

Study objective:

This study wants to investigate the direct effects of intramuscular testosterone replacement versus placebo in changing the intrahepatic fat content, myocardial fat content, visceral and abdominal fat content as well as pancreatic fat content of poorly controlled men suffering from T2DM and secondary hypogonadism. Furthermore, the effects of testosterone on glycaemic control and cardiovascular safety will be investigated. The effect of testosterone on cardiac perfusion will be tested in this high risk collective.

For studying long-term effects, an open-label extension of the study by an additional 2 years is intended.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes/T2DM
* male sex
* HbA1c >=5.7% -9.0% or fasting glucose >=100mg/dl or postprandial glucose>= 140mg/dl
* Age >=18 -75 years
* BMI>=25kg/m²
* Hypogonadism assessed by laboratory testing (testosterone < 4,04ng/ml (=14nmol/l) Metformin 8 weeks stable dose, SGLT2 inhibitors 3 months stable dose, DPP4 inhibitors 3 months stable dose, GLP1 RA 3 months stable dose and long acting insulin (basal insulin) 8 weeks stable dose
* able and willing to not change diet and physical activity during enrollment in study
* consent and able to give informed consent.

Exclusion Criteria:

* Current testosterone treatment or testosterone replacement within the last 12 month
* Serum creatinine>1,5mg/dl
* Liver enzymes above 3 fold normal range
* PSA>4.0μg/l
* Hematocrit>50%
* Known intolerance to testosterone undecanoate or any of its ingredients
* Myocardial infarction within the last 12month
* Stroke within the last 12 month
* Untreated congestive heart disease
* malignancy within the last 5 years before randomization
* Prostate cancer or any suspicion thereof
* Breast cancer
* Liver tumor/cancer
* Epilepsy
* Migraine
* Presence of any absolute or relative contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* patients on antidiabetic medication like Sulfonylurea or Glitazones.
* Any other clinical condition that would jeopardize patients safety while participating in this clinical trial
* Known autoimmune disease or chronic inflammatory condition
* Other liver disease including chronic viral hepatitis (B or C), alcohol abuse, hemochromatosis, alpha-1 antitrypsin deficiency, autoimmune hepatitis, Wilson's disease, primary sclerosing cholangitis or primary biliary cirrhosis, or liver cirrhosis of any etiology
* Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
* History of bariatric surgery
* Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight
* Subjects receiving antihypertensive medication and/or thyroid hormones, the dose(s) of which have not been stable for at least 6 weeks prior to baseline
* Uncontrolled/ untreated hypertension
* Current treatment with systemic steroids at time of informed consent. (Treatment with local and inhaled steroids is allowed)
* Donation of blood (> 400 mL) during the previous 3 months prior to the screening visit or during the duration of the study
* Participation in another trial with an investigational drug within 30 days prior to informed consent.
* Pharmacist, study coordinator, other staff thereof, directly involved in the conduct of the protocol.
* contraindication for intramuscular injection (e.g patient receiving anticoagulants on a regular basis such as NOAKs or VKAs, or DAPT).
* COPD Gold IV or recurrent acute or allergic asthma (for MPI)
* Contraindications for cardiac stress test as acute myocardial infarction, instable angina, severe hypertension, myocarditis, life threatening rhythmic disorders without physical activity.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Liver fat | baseline to week 52, and after 2 years follow up
  Change in Liver fat content

SECONDARY OUTCOMES:
body weight | baseline to week 52, and after 2 years follow up
  change in body weight
waist, hip and neck circumference | baseline to week 52, and after 2 years follow up
  change in waist, hip and neck circumference
insulin sensitivity | baseline to week 52, and after 2 years follow up
  change in insulin sensitivity and Insulin secretion assessed by oGTT
Level of HbA1c | baseline to week 52, and after 2 years follow up
  change in HbA1c from baseline to week 52
Concentration of lipids | baseline to week 52, and after 2 years follow up
  change in lipid profile from baseline and free fatty acids in the OGTT
quality of live questionnaire | baseline to week 52, and after 2 years follow up
  change of quality of live assessed by WHO 5 Well Being Questionnaire
blood pressure | baseline to week 52, and after 2 years follow up
  change in systolic and diastolic blood pressure
sexual function questionnaire | baseline to week 52, and after 2 years follow up
  change sexual function assessed by International Index of Erectile Dysfunction questionnaire
diabetes management satisfaction questionnaire | baseline to week 52, and after 2 years follow up
  change of diabetes management satisfaction assessed by Diabetes Treatment Satisfaction Questionnaire

OTHER OUTCOMES:
amount of body fat | baseline to week 52, and after 2 years follow up
  Change in body fat, liver volume, visceral adipose tissue, subcutaneous adipose tissue, total adipose tissue and total lean tissue, myocardial and pancreatic fat and ventricular function
level of HbA1c | baseline to week 52, and after 2 years follow up
  The occurrence of treat to target efficacy i.e. HbA1c < 7.0 % or < 6.5 %.
HbA1c reduction >=0.5% | baseline to week 52, and after 2 years follow up
  The occurrence of a relative efficacy response. i.e. HbA1c lowering of at least 0.5%
mean daily glucose profile | baseline to week 52, and after 2 years follow up
  The change from baseline in mean daily glucose profile assessed by 8 point glucose profiles
weight | baseline to week 52, and after 2 years follow up
  The change in weight (>5% and >10%)
IMT | baseline to week 52, and after 2 years follow up
  Change in Intima Media Thickness
Albumin/ Creatinine Ratio | baseline to week 52, and after 2 years follow up
  Change in Albumin/ Creatinine Ratio
myocardial flow reserve | baseline to week 52, and after 2 years follow up
  Change in myocardial flow reserve
concentration of osteocalcin | baseline to week 52, and after 2 years follow up
  Change in concentration of osteocalcin
amount of visceral adipose tissue, | baseline to week 52, and after 2 years follow up
  Change in amount of visceral adipose tissue,
amount of subcutaneous adipose tissue, | baseline to week 52, and after 2 years follow up
  change in amount of subcutaneous adipose tissue,
amount of total lean tissue, | baseline to week 52, and after 2 years follow up
  change in amount of total lean tissue,
amount of myocardial fat | baseline to week 52, and after 2 years follow up
  change in amount of myocardial fat
amount of pancreatic fat | baseline to week 52, and after 2 years follow up
  change in amount of myocardial fat

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, MD, Principal Investigator — Medical University Vienna; Jürgen Harreiter, PhD, Principal Investigator — Medical University Vienna
Locations (1):
- Abt. für Endokrinologie & Stoffwechsel, Univ. Klin f. Innere Medizin III, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Individual data that underlie the results reported in this article, after deidentification of this
Supporting Information: Study Protocol
Time Frame: beginning 6 months and ending 24 months following article publication
Access Criteria: Researches who provide a methodologically sound proposal. Please send the proposal to juergen.harreiter@meduniwien.ac.at. A data access agreement needs to be signed.